CLINICAL TRIAL: NCT05595174
Title: Assessment of Maxillary Canine Retraction Using Self-ligating Brackets System Assisted With Micro-osteoperforations: A Prospective Controlled Clinical Study
Brief Title: Assessment of Maxillary Canine Retraction Using Self-ligating Brackets System Assisted With Micro-osteoperforations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Khaled Sobhy Abdelaziz, doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 850/2057
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Accerleration of Tooth Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): Patient with self-ligating bracket system split mouth with and without micro-osteoperforations.
  Extraction of first premolars were done. A standardized wire sequence of .012'', 0.014'',0,016'', and 0.016''×0.022'' nickel-titanium were followed to achieve leveling and alignment.
  Interventions: Biological: self ligating bracket with micro osteoperforation; Biological: self ligating bracket without micro osteoperforation
- group 2 (Active Comparator): Patient with conventional bracket with split mouth with and without micro-osteoperforations.
  Extraction of first premolars were done. A standardized wire sequence of .012'', 0.014'',0,016'', and 0.016''×0.022'' nickel-titanium were followed to achieve leveling and alignment.
  Interventions: Biological: conventional bracket with micro osteoperforation; Biological: conventional bracket without micro osteoperforation

INTERVENTIONS:
Biological: self ligating bracket with micro osteoperforation — A standardized wire sequence of .012'', 0.014'',0,016'', and 0.016''×0.022'' nickel-titanium were followed to achieve leveling and alignment. Micro-osteoperforations will be formed
  Arms: group 1
Biological: conventional bracket with micro osteoperforation — A standardized wire sequence of .012'', 0.014'',0,016'', and 0.016''×0.022'' nickel-titanium were followed to achieve leveling and alignment. Micro-osteoperforations will be formed.
  Arms: group 2
Biological: conventional bracket without micro osteoperforation — A standardized wire sequence of .012'', 0.014'',0,016'', and 0.016''×0.022'' nickel titanium were followed to achieve leveling and alignment
  Arms: group 2
Biological: self ligating bracket without micro osteoperforation — A standardized wire sequence of .012'', 0.014'',0,016'', and 0.016''×0.022'' nickel-titanium were followed to achieve leveling and alignment.
  Arms: group 1

SUMMARY:
Assessment of maxillary canine retraction using self-ligating brackets system assisted with micro-osteoperforations: A prospective controlled clinical study

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients between the age (14-20 y).
* Patients indicated for maxillary first premolar extraction.
* Angle's Class I bimaxillary, Class II Division 1 malocclusion (ANB <5).
* Irregularity index < 4 mm.
* No previous orthodontic treatment.
* Fully erupted dentition.

Exclusion Criteria:

* Patients not indicated for non-extraction approach.
* Prominent canine root (in labial cortical bone).
* History of systemic and medical illness that could interfere with OTM.
* Previous orthodontic treatment.
* Extreme skeletal class II occlusion (ANB >5).
* Poor oral hygiene or periodontally compromised patient

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
effect of canine retraction | at 6 months
  assessment of maxillary canine retraction rate using self-ligating brackets system assisted with micro-osteoperforations.

CONTACTS AND LOCATIONS:
Overall Officials: khaled sobhy abdelaziz, master, Principal Investigator — Al-Azhar University
Locations (1):
- Alazhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Abbing A, Koretsi V, Eliades T, Papageorgiou SN. Duration of orthodontic treatment with fixed appliances in adolescents and adults: a systematic review with meta-analysis. Prog Orthod. 2020 Oct 5;21(1):37. doi: 10.1186/s40510-020-00334-4. PMID 33015719